CLINICAL TRIAL: NCT05510739
Title: Support for Physical Activity in Everyday Life With Parkinson's Disease Using eHealth Technology
Brief Title: Support for Physical Activity in Everyday Life With Parkinson's Disease
Acronym: STEPS-PD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stiftelsen Stockholms Sjukhem (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: StockholmsSjukhem
Record Dates: First submitted 2022-07-25; First posted 2022-08-22 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease; Physical Activity; eHealth; Gait Disorders, Neurologic
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motor-cognitive exercise using eHealth (Experimental): 10-week eHealth based motor-cognitive home training using digital tablets. Cognitive behavioural strategies to promote increase in physical activity levels (walking). Participants will be encouraged to perform 150 minutes of home exercise per week, occurring on three non-consecutive days.
  Interventions: Behavioral: Motor-cognitive home exercise supported by eHealth technology
- Individualised home training program (Active Comparator): Participants will receive an individualized home exercise program on paper and one instructional session. They will receive written instructions on performing the program 2-3 times weekly and instructions on exercise progression. They will receive no support during the 10-week period.
  Interventions: Behavioral: Individualized home exercise program

INTERVENTIONS:
Behavioral: Motor-cognitive home exercise supported by eHealth technology — 10-week, individualized and progressive exercise program targeting functional strength, cardiovascular fitness and physical activity levels. Cognitive exercises are incorporated with motor exercises as an adjunct to the intervention.
  Arms: Motor-cognitive exercise using eHealth
Behavioral: Individualized home exercise program — Individualised home exercise program leaflet involving one initial instruction session. Written instructions involving dose and exercise progression. No support during the 10 week period.
  Arms: Individualised home training program

SUMMARY:
This study aims to determine the effects of a motor-cognitive exercise intervention, delivered in the home environment using eHealth methods, among people with Parkinson's disease. The intervention will support and motivate motor training, combined with cognitive training, aimed at attentional and executive functions, among people at mild-moderate disease stages. The main hypothesis is that unsupervised motor-cognitive training in the home environment using eHealth will lead to improvements in gait performance, increased physical activity levels and improved perceived health.

DETAILED DESCRIPTION:
This randomised controlled trial will investigate the efficacy of a motor-cognitive exercise program in the home environment, over a 10-week period, on physical function, and motor-cognitive dual task function as well as physical activity behavior in everyday life. A follow-up assessment comprising health-related questionnaires and physical activity monitoring will be conducted at one year post-intervention. Participants will be recruited through Stockholms sjukhem foundation, Karolinska University and via announcements in relevant forums like for instance the Swedish Parkinson Association. Consenting participants will be randomized to the eHealth Intervention group or the control group condition. Block randomization will be achieved using a computerized random sequence generator. Blinded assessors will perform the pre- and post-intervention testing of physical performance.

The ultimate aim of this project is to provide people with PD with continual long-term and evidence-based rehabilitation in their everyday lives using mobile health technology, to support their self- management and increase their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson´s disease
* Hoehn & Yahr (Parkinsons progression scale) 2-3
* ≥ 50 years of age
* Able to ambulate indoors without mobility aid
* Able to walk continually with/without a walking aid for at least 6 minutes

Exclusion Criteria:

* Cognitive impairment affecting the ability to understand or follow verbal or written instructions (Montreal Cognitive Assessment ≤ 21 points
* Major problems with freezing and/or two or more falls in the month previous to inclusion
* Other existing neurological/ orthopedic or cardiovascular disease which impedes the performance of unsupervised exercise
* Impaired vision and/or impaired communication which hinders participation
* No internet connection in the home

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The six minute walk test | Change in balance performance at 10 weeks
  This test measures walking capacity by measuring the distance covered (meters) over a time period of 6 minutes.

SECONDARY OUTCOMES:
Gait parameters during single and dual-task conditions | Change at 10 weeks
  Stride length (meters); Cadence (steps/ minute) will be captured using born-worn inertial sensors
Quality of life questionnaires | Change at 10 weeks and one year post-intervention
  PDQ-39 is disease specific quality of life questionnaire. Items are grouped into eight scales that are scored by expressing summed item scores as a percentage score ranging between 0 and 100
Physical activity measured with accelerometers | Change at 10 weeks and one year post-intervention
  Steps per day and time (minutes) in different physical activity intensities (high,moderate and low intensity)
Dual-task ability during walking | Change at 10 weeks
  Captured using the Auditory Stroop test during walking and expressed as percentage error of the task
Balance ability | Change at 10 weeks
  MiniBest test. Scoring 0-28, lower scores = greater balance impairment
Executive function | Change at 10 weeks
  Trail making test A & B. Expressed as time required to perform the test (seconds)
Balance Confidence | Change at 10 weeks and one year post-intervention
  The Activities-specific Balance Confidence scale is a measure of confidence performing in various activities without losing balance or experiencing unsteadiness. A 16-item self-report measure with items rated on a rating scale that ranges from 0-100. A higher score indicates higher balance confidence.
Health-related Quality of Life | Change at 10 weeks and one year post-intervention
  The EQ-5D is a two-part instrument that measures health-related quality of life. It examines 5 domains of quality of life: mobility, self-care, daily activities, pain, anxiety/depression. It comprises 5 questions and a visual scale.
Exercise Self-Efficacy | Change at 10 weeks and one year post-intervention
  The Exercise Self-Efficacy Scale is an instrument examining confidence regarding carrying out regular physical activities and exercise. Questions are answered on a 4-point rating scale. A higher score indicates greater confidence.
Walking ability | Change at 10 weeks and one year post-intervention
  The Walk-12 questionnaire examines limitations in walking ability. It consists of 12 questions answered on either a 3-point or 5-point rating scale.
Hospital Anxiety and Depression Scale | Change at 10 weeks and one year post-intervention
  A 14-item measure designed to reflect the state of generalised anxiety and depression. The respondent rates each item on a 4-point scale. Higher scores indicate greater levels of anxiety or depression.
Life Space Assessment | Change at 10 weeks and one year post-intervention in only the final cohort of participants
  The LSA is a self-report measure of the frequency of independent mobility across 5 life-space levels. Higher scores indicate more life-space and movement throughout the community.
Global Positioning System | Change at 10 weeks and one year post-intervention in only the final cohort of participants
  GPS monitors collecting participant daily location and movement data via latitude and longitude coordinates collected throughout waking hours.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ankarcrona, PhD, Study Chair — Karolinska Institutet, NVS; Sofia Pettersson, MSc, Study Chair — Stockholms Sjukhem Foundation, Primary Care Rehabilitation
Locations (1):
- Stockholms sjukhem, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Currently we do not have IRB for sharing

REFERENCES:
- [Derived] Leavy B, Sedhed J, Kalbe E, Akesson E, Franzen E, Johansson H. Design of the STEPS trial: a phase II randomized controlled trial evaluating eHealth-supported motor-cognitive home training for Parkinson's disease. BMC Neurol. 2023 Oct 4;23(1):356. doi: 10.1186/s12883-023-03389-y. PMID 37794320